CLINICAL TRIAL: NCT03778255
Title: Comparing the Diagnostic Value of Different Lymph Node Tracing Methods in Detecting Sentinel Lymph Node Metastasis in Endometrial Cancer
Brief Title: Sentinel Lymph Node Mapping In Endometrial Cancer
Acronym: SLNMIEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Peking University International Hospital (Other); Shanghai First Maternity and Infant Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Sun Yat-sen University (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); Cancer Hospital of Guangxi Medical University (Other); First People's Hospital of Foshan (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Affiliated Hospital of Zhengzhou University (Other); Beijing Blue Sky Shared Health Management Co., Ltd. (Unknown); Chongqing Lummy Pharmaceutical Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018PHD002-01
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Endometrial Neoplasms
Keywords: Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: The procedure is listed as follows:
  1. Recruiting endometrial cancer patients undergoing hysterectomy with or without bilateral adnexectomy, pelvic and para-aortic lymph node resection from July 2018 to June 2020.
  2. Selecting the Standard-compliant patients according to the inclusion and exclusion criteria and letting them sign an informed consent form.
  3. Numbering the above patients and collecting their clinical data.
  4. Injecting carbon nanoparticles (CNP)[Not Equipped with near-infrared fluorescent vascular imager] or CNP combining Indocyanine Green(ICG)[Equipped with near-infrared fluorescent vascular imager].
  5. Identifying and removing sentinel lymph nodes.
  6. Completing the hysterectomy with or without bilateral adnexectomy, pelvic and para-aortic lymph node resection
  7. Staining all nodes using hematoxylin-eosin staining.
  8. Calculating the sensitivity, negative predictive value, etc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Undergoing sentinel lymph node biopsy (Experimental)
  Interventions: Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — 1. Injecting carbon nanoparticles (CNP)[Not Equipped with near-infrared fluorescent vascular imager] or CNP combining Indocyanine Green(ICG)[Equipped with near-infrared fluorescent vascular imager].
  2. Identifying and removing sentinel lymph nodes.
  3. Staining all nodes using hematoxylin-eosin staining.

SUMMARY:
Lymph node assessment provides the crucial information about the prognosis of endometrial cancer. Sentinel lymph node stands in the first station on the lymph node metastasis pathways. While traditional systemically lymph node resection would bring a lot of complications, sentinel node mapping and biopsy is a feasible way with less damage to evaluate whether lymph node metastasis occurs in endometrial cancer patients, due to less lymph nodes resected. However, the process of this technology in endometrial cancer isn't well established. The investigators intend to conduct a prospective and multicentric study to evaluate the effectiveness of different mapping methods to achieve a reliable lymph node assessment. Endometrial cancer patients in each center will be recruited in the investigators' study with inclusion and exclusion criteria. After the patients signing the informed consent form, the surgery process will be performed, including sentinel lymph node mapping with Carbon Nanoparticles (CNP) or CNP combining Indocyanine Green(ICG), hysterectomy with or without bilateral adnexectomy, pelvic and para-aortic lymph node resection, sequentially. All resected nodes will be pathologically exanimated. Then the data obtained will be analyzed and discussed deeply and finally lead to a conclusion.

DETAILED DESCRIPTION:
Quality Control The investigators' quality assurance plan is as follows. A. Once the plan has been approved, it cannot be modified at will. If special circumstances such as difficulty in implementation are found after the start of the study, the proposal may be revised or supplemented by the discussion of the research group and the project leader, and the revised content shall be recorded in writing.

The program change process is as follows:

* Identify the problems and understand the necessary to change the plan;
* Convene the main members of the research team and the project leader to discuss and propose solutions;
* Revise the plan and update the version number, fill out the "Program Description";
* The revised plan and the "Revision of the Plan" need to be signed by the person in charge of the project. If necessary, they must be submitted to the ethics committee for approval or filing; if approved, the revised plan can be implemented.

B. In order to ensure that the research personnel have sufficient qualifications to undertake specific research work, the research personnel should at least complete the following training before the project starts:

* Research object protection and ethical requirements;
* Study protocols and related standard operating procedures (tracer injection methods, use of near-infrared fluorescent vascular imagers, and pathology);
* Case Report Form and gauge filling instructions (form entry criteria, surgical record methods, etc.);
* Clinical research project implementation considerations (such as research object screening, enrollment, data collection process); Project-related training should be carried out throughout the research process. The project leader and project coordinator can increase the training content according to the situation, such as training on weak links in the test, training on updating programs and various causes.

Data Management A. Case report form design The researcher is responsible for drafting the research case report form. B. Data Entry and Data Verification According to the final version of CRF, the project database is built using software. The data entry and verification is carried out by a dedicated person.

Statistical Analysis A. Statistical Analysis Plan and Statistical Software After the trial protocol is determined, the statistical professors and the main investigators are responsible for developing a statistical analysis plan. The statistical analysis software uses SAS® 9.2 software (software installation point authorization number: 11202165).

B. Calculation and reasoning of sample size The sample size is calculated using PASS11 software; the sample size is estimated based on the negative prediction value of the previous study, and the negative prediction value of SLNs is expected to be 95%; the allowable error is 2% (the range of the confidence interval is 93% to 97%). When the significant level is 0.05, 508 cases are needed to be studied. Considering the detection rate of 80% of SLNs, a total of 635 cases are expected to be studied.

C. Statistical Analysis Methods General principle Using a two-sided test, a P value of less than 0.05 would be considered statistically significant.

The quantitative indicators will calculate the mean, standard deviation, median, minimum, maximum, lower quartile (Q1), upper quartile (Q3), and the classification indicators will describe the number of cases and percentages.

Comparison of clinicopathological features (age, body mass index, pathological type, tumor stage, grading, maximum tumor diameter, invasive myometrial depth, lymphatic vascular infiltration, and tracer method) for SLNs and undetected SLNs will be based on the type of indicator. For the comparison of quantitative data between groups, the t-test or Wilcoxon rank sum test will be used according to the data distribution. For the comparison of categorical data between groups, the data will be analyzed by chi-square test or exact probability method (if the chi-square test is not applicable). And the grade data was analyzed by Wilcoxon rank sum test or CMH test.

Clinical diagnostic index calculation According to the true positive (TP), false negative (FN), true negative (TN), and false positive (FP), the results of SLNs pathological examination and all lymph node pathological examination results will be compared. The comparison results will be plotted as a four-grid table to calculate sensitivity, false negative rate, and negative predictive value, respectively.

Chi-square test or exact probability method (if the chi-square test is not applicable) will be used to compare the clinical diagnosis value of SLNs biopsy of endometrial cancer patients with injection of carbon nanoparticles (CNP) or combined injection of CNP and indocyanine green(ICG).

Chi-square test or exact probability method (if the chi-square test is not applicable) will be used to analyze the clinic-pathological factors affecting the detection rate of SLNs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometrial cancer (including all pathological type and clinical stage).
* Decide to receive hysterectomy with or without bilateral adnexectomy, pelvic and para-aortic lymph node resection
* Agree to conduct the study and sign an informed consent form

Exclusion Criteria:

* History of previous pelvic or inguinal lymphadenectomy or other history of surgery affecting the uterine lymphatic drainage
* Other history of pelvic or abdominal malignant tumors in the past 5 years
* Intolerable for surgery due to severe comorbidities
* During a period of pregnancy
* Allergic to the tracer
* Diagnosis of uncontrolled epilepsy, central nervous system disease or mental disorder, with the judgment from the investigator that the above diseases would affect clinical research compliance.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value | Through study completion, an average of 2 years
  Sentinel lymph node detection is defined as at least one lymph node is found in a patient. Sentinel lymph node negative is defined as no sentinel lymph node detected. True negative is defined as no metastasis found in both sentinel lymph nodes (SLNs) and non-SLNs. Negative predictive value is defined as the proportion of true negative patients to SLNs negative patients in patients with sentinel lymph nodes detected, which means patients without SLNs detected won't be included in the calculation.

SECONDARY OUTCOMES:
detection rate | Through study completion, an average of 2 years
  Sentinel lymph node detection is defined as at least one lymph node is found in a patient. The detection rate is the proportion of the patients with SLNs detected in all enrolled patients.
Sensitivity | Through study completion, an average of 2 years
  Sensitivity is defined as the proportion of the SLNs positive patients in patients with SLNs or non-SLNs lymphatic metastasis (among the patients with SLNs detected)
False negative rate | Through study completion, an average of 2 years
  False negative is defined as no metastasis found in SLNs while metastasis found in non-SLNs. False negative rate is defined as the proportion of the false negative patients in the patients with SLNs or non-SLNs lymphatic metastasis(among the patients with SLNs detected)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hosoital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Creasman WT, Morrow CP, Bundy BN, Homesley HD, Graham JE, Heller PB. Surgical pathologic spread patterns of endometrial cancer. A Gynecologic Oncology Group Study. Cancer. 1987 Oct 15;60(8 Suppl):2035-41. doi: 10.1002/1097-0142(19901015)60:8+3.0.co;2-8. PMID 3652025
- [Background] May K, Bryant A, Dickinson HO, Kehoe S, Morrison J. Lymphadenectomy for the management of endometrial cancer. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007585. doi: 10.1002/14651858.CD007585.pub2. PMID 20091639
- [Background] Benedetti Panici P, Basile S, Maneschi F, Alberto Lissoni A, Signorelli M, Scambia G, Angioli R, Tateo S, Mangili G, Katsaros D, Garozzo G, Campagnutta E, Donadello N, Greggi S, Melpignano M, Raspagliesi F, Ragni N, Cormio G, Grassi R, Franchi M, Giannarelli D, Fossati R, Torri V, Amoroso M, Croce C, Mangioni C. Systematic pelvic lymphadenectomy vs. no lymphadenectomy in early-stage endometrial carcinoma: randomized clinical trial. J Natl Cancer Inst. 2008 Dec 3;100(23):1707-16. doi: 10.1093/jnci/djn397. Epub 2008 Nov 25. PMID 19033573
- [Background] ASTEC study group; Kitchener H, Swart AM, Qian Q, Amos C, Parmar MK. Efficacy of systematic pelvic lymphadenectomy in endometrial cancer (MRC ASTEC trial): a randomised study. Lancet. 2009 Jan 10;373(9658):125-36. doi: 10.1016/S0140-6736(08)61766-3. Epub 2008 Dec 16. PMID 19070889
- [Background] Todo Y, Kato H, Kaneuchi M, Watari H, Takeda M, Sakuragi N. Survival effect of para-aortic lymphadenectomy in endometrial cancer (SEPAL study): a retrospective cohort analysis. Lancet. 2010 Apr 3;375(9721):1165-72. doi: 10.1016/S0140-6736(09)62002-X. Epub 2010 Feb 24. PMID 20188410
- [Background] NCCN Guidelines Version 1. 2018. Uterine Neoplasms [EB/OL]. [2018-02-10]. http://www.nccn.org/professionals/physician_gls/pdf/uterine.pdf.
- [Background] Lu Y, Wei JY, Yao DS, Pan ZM, Yao Y. Application of carbon nanoparticles in laparoscopic sentinel lymph node detection in patients with early-stage cervical cancer. PLoS One. 2017 Sep 5;12(9):e0183834. doi: 10.1371/journal.pone.0183834. eCollection 2017. PMID 28873443
- [Background] Holloway RW, Abu-Rustum NR, Backes FJ, Boggess JF, Gotlieb WH, Jeffrey Lowery W, Rossi EC, Tanner EJ, Wolsky RJ. Sentinel lymph node mapping and staging in endometrial cancer: A Society of Gynecologic Oncology literature review with consensus recommendations. Gynecol Oncol. 2017 Aug;146(2):405-415. doi: 10.1016/j.ygyno.2017.05.027. Epub 2017 May 28. PMID 28566221
- [Background] Liang SC, Wang ZQ, Wang JL. [Clinical analysis of 76 cases of sentinel lymph node detection in cervical cancer and endometrial cancer]. Zhonghua Fu Chan Ke Za Zhi. 2017 Sep 25;52(9):605-611. doi: 10.3760/cma.j.issn.0529-567X.2017.09.006. Chinese. PMID 28954449